CLINICAL TRIAL: NCT02328378
Title: Postoperative Pain Relief After Cesarean Section: Is There a Role for the Quadratus Lumborum Block?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Tarek Ansari (Other)
Responsible Party: Sponsor-Investigator, Dr. Tarek Ansari, Consultant Anesthetist, Corniche Hospital
Organization: Corniche Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ch27021403
Record Dates: First submitted 2014-12-25; First posted 2014-12-31 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quadratus Lumborum block group (QL) (Active Comparator): patients will receive a bilateral Quadratus Lumborum block using Bupivicaine 0.125%
  Interventions: Procedure: Quadratus Lumborum block
- Control Group (Placebo Comparator): patients will receive a bilateral placebo block
  Interventions: Procedure: Quadratus Lumborum block

INTERVENTIONS:
Procedure: Quadratus Lumborum block — Patients will receive a bilateral Quadratus Lumborum block using 0.125% Bupivacaine in a dose of 0.2ml/kg body weight, after the end of surgery.

SUMMARY:
The Quadratus Lumborum block (QLB) was first described by Blanco in 2007. The main advantage of QLB compared to the Transversus Abdominis Plane block (TAP) is the extension of local anesthetic agent beyond the TAP plane to the thoracic paravertebral space. The wider spread of the local anesthetic agents produces extensive analgesia and prolonged action of the injected local anesthetic solution.

Previous studies showed that TAP block may not be effective in improving postoperative analgesia in patients who had cesarean section under spinal anaesthesia.

The aim of this randomised controlled, double blinded study is to examine the effect of QLB on the postoperative pain management in patients who had cesarean section under spinal anesthesia.

DETAILED DESCRIPTION:
After ethical committee approval, informed written consent will be obtained from all patients. A Sample size of 25 patients per group was calculated based on 15% reduction in morphine consumption with 0.05% significance and a power of 0.8.

Consenting patients scheduled to have elective cesarean section under spinal anesthesia will be randomised to undergo QLB with Bupivacaine versus placebo(saline) after their surgery. Allocation will be done using closed envelope technique.

The study medications/placebo will be prepared and labelled by an anesthetist who is not involved in the study.

All patients will receive a standard spinal anesthetic. At the end of surgery , Quadratus lumborum block group (QL) patients will receive bilateral QLB with 0.125% bupivacaine.

Control group patients will receive a bilateral placebo block using saline. The block will be performed in operation theatre after the end of cesarean section with intravenous access, ECG, BP, oxygen saturation by pulse oximetry monitoring and full resuscitation equipment and medication ready.

The patient will be placed in a lateral position with the side to be blocked facing upwards. The ultrasound probe will be properly sterilized and with sterile covers.

A 22 Gauge, two inch Pajunk Sonoplex needle is advanced under ultrasound guidance on the posterior aspect of the Quadratus Lumborum. Following negative aspiration, 0.2 ml/kg of 0.125% bupivacaine, or placebo(saline) is injected in each side with intermittent aspiration and the spread of injectate followed on ultrasound.

All patients will receive the routine postoperative analgesia, comprising patient-controlled IV morphine analgesia and regular diclofenac and paracetamol.

All patients will be assessed postoperatively by a blinded investigator: in the postanesthesia care unit and at 2, 4, 6, 12, 24, 36, and 48 h postoperatively

ELIGIBILITY:
Inclusion Criteria:

* Elective caesarean sections
* ASA 1 to 3
* Written informed consent.

Exclusion Criteria:

* Patient refusal
* Local infection at the site of injection
* Allergy to study medications
* Sepsis
* Anatomic abnormalities
* Systemic anticoagulation or coagulopathy
* Inability to comprehend or participate in pain scoring system
* Inability to use intravenous patient controlled analgesia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Total morphine used in the first 48 hours after surgery | 48 hours
  Total cumulative morphine dose in mg used in the first 48 hours after surgery

SECONDARY OUTCOMES:
Nausea or vomiting | 48 hours
  Categorical assessment of nausea. 0 = No Nausea
  1. = Mild Nausea.
  2. = Moderate
  3. = Severe Nausea or Vomit
Sedation score in the first 48 hours | 48 hours
  Categorical assessment of sedation. 0 = wide awake
  1. = drowsy but responds to normal verbal communication.
  2. = asleep, but awakes with verbal communication.
  3. = asleep, awakens with mild physical stimulation.
  4. = asleep, unresponsive to mild physical stimulation.
Severity of postoperative pain via visual analogue pain scale | 48 hours
  VAS range from 0 for no pain to 10 for worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Rafa Blanco, FRCA, Principal Investigator — Corniche Hospital; Tarek Ansari, FFARCSI, Principal Investigator — Corniche Hospital; Emad Girgis, MD, Principal Investigator — Corniche Hospital
Locations (1):
- Corniche Hospital, Abu Dhabi, United Arab Emirates

REFERENCES:
- [Derived] Blanco R, Ansari T, Girgis E. Quadratus lumborum block for postoperative pain after caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2015 Nov;32(11):812-8. doi: 10.1097/EJA.0000000000000299. PMID 26225500